CLINICAL TRIAL: NCT01228045
Title: A Phase 2 Study of Trastuzumab in Combination With TS-ONE and Cisplatin in First-line Human Epidermal Growth Factor Receptor 2 (HER2)-Positive Advanced Gastric Cancer.
Brief Title: A Study of Trastuzumab in Combination With TS-ONE & Cisplatin in First-line Human Epidermal Growth Factor Receptor 2 (HER2)-Positive Advanced Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National Cancer Centre, Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S1/CDDP/Her
Record Dates: First submitted 2010-10-21; First posted 2010-10-25 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-06

CONDITIONS: Gastric Cancer
Keywords: Patients with histologically proved adenocarcinoma of advanced gastric cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Trastuzumab; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Trastuzumab in Combination with TS-ONE and cisplatin (Experimental): The initial dose of cisplatin is fixed to be 60 mg/m2 and intravenously administered over 1 hour on day 1 of the cycle. TS-ONE is orally administered consecutive 14-day followed by 7-day rest. The initial standard dose of TS-ONE is determined based on the body surface area tabled below. Trastuzumab is intravenously administered with the loading dose of 8 mg/kg followed by maintenance dose of 6mg/kg in day 1 of each cycle. The study treatments are repeated every 3 weeks. Study treatment can continue until PD, but cisplatin can be skipped or discontinued if patients experienced unbearable toxicity which comes from cisplatin.
  Interventions: Drug: Trastuzumab in Combination with TS-ONE and cisplatin

INTERVENTIONS:
Drug: Trastuzumab in Combination with TS-ONE and cisplatin — Subjects will receive treatment that combined TS-ONE, cisplatin and trastuzumab every 3 weeks in this study. This 3 weeks period of time is called a cycle. The cycle will be repeated until subject experience disease progression or unbearable toxicities or they choose to withdraw from the study. Each cycle is numbered in order.

SUMMARY:
The investigators hypothesis is that the combination of TS-ONE with cisplatin and trastuzumab is safe and as effective as combination treatment for HER2 positive gastric cancer.

DETAILED DESCRIPTION:
Gastric carcinoma is the second most common cause of cancer death world-wide. Approximately 875,000 patients are diagnosed world-wide with gastric cancer each year. Gastric cancer is often diagnosed at an advanced stage1. At diagnosis, while some patients have gastric carcinoma that extends within loco-regional confines and can undergo a curative resection, many patients cannot undergo curative resection. Gastric cancer continues to pose a major medical challenge.

While advanced gastric carcinoma is incurable, chemotherapy can have a palliative effect in symptomatic patients. Chemotherapy improves outcome compared to best supportive care in gastric cancer. Various chemotherapeutic agents including 5-FU, mitomycin, etoposide, cisplatin, irinotecan and the taxanes, have demonstrated activity as monotherapy. Combination chemotherapy has been shown to have better survival outcomes than single agent chemotherapy Standard chemotherapy for advanced gastric carcinoma includes a fluoropyrimidine and platinum -based combination chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically proved adenocarcinoma of advanced gastric cancer.
2. Patients who have HER2-positive cancer confirmed with IHC and/or FISH.
3. Patients with proved presence of measurable (RECIST criteria) lesions within 28 days before enrollment.
4. Patients without prior treatment (ex. radiotherapy, chemotherapy, hormonal therapy): Patients who completed adjuvant chemotherapy more than 180 days before may be enrolled but those who received TS-ONE or cisplatin shall be excluded.
5. Patients with the following function of bone marrow, liver and kidney based on the laboratory tests measured within 14 days before enrollment. Hemoglobin >= 8.0 g/dL leukocytes >=3,000/mcL absolute neutrophil count >=1,500/mcL platelets >=100,000/mcL total bilirubin within normal institutional limits AST(SGOT)/ALT(SGPT)=<2.5 X institutional upper limit of normal ALP < twice of the upper limit of normal, creatinine within normal institutional limits or creatinine clearance >=60 mL/min for patients with creatinine levels above institutional normal (When AST(GOT), ALT(GPT) and ALP do not satisfy the conditions above and these values are considered to be caused by cancer, the decision is based on the discretion of investigators or co-investigators) Creatinine clearance can be estimated using Cockcroft-Gault formula man: Ccr (mL/min) = body weight (kg) x (140 - age)/(72 x serum creatinine (mg/dL)), woman: Ccr = male Ccr x 0.85].
6. ECOG performance status =<2 (Karnofsky >60%; see Appendix A).
7. Patients who are expected to survive more than 3 months after enrollment.
8. Age >= 21.
9. Patients of adequate oral intake.
10. Patients who underwent electrocardiography within 28 days before enrollment.\
11. Patients who give written informed consent for additional endoscopy to obtain fresh frozen tissue biopsies for translational studies at 2 time points pre-1st cycle of chemotherapy and at progression.
12. Patients who give written informed consent for enrollment into trial.

Exclusion Criteria:

1. Patients for whom TS-ONE or cisplatin or trastuzumab is contraindicated.
2. History of allergic reactions attributed to compounds of similar chemical or biologic composition to TS-ONE, cisplatin and trastuzumab.
3. Patients receiving any other investigational agents.
4. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
5. Baseline heart function LVEF (Left Ventricular Ejection Fraction) < 50%.
6. Patients with serious (ex. inpatient care is needed) complications (ex. intestinal paralysis, intestinal occlusion, interstitial pneumonia or pulmonary fibrosis, poorly-controlled diabetes, renal failure or hepatic cirrhosis).
7. Patients with massive ascites (moderate or higher, beyond the pelvic cavity and retention on the anterior surface of the liver on CT) or pleural effusion retention.
8. Patients with extensive bone metastasis.
9. Patients with known brain metastases.
10. Patients with fresh bleeding from the digestive tract which needs repeated blood transfusion.
11. Patients with diarrhea (4 or more times per day or watery diarrhea).
12. Patients with simultaneously active multiple cancer.
13. Pregnant or lactating female.
14. Patients with reproductive potential who refuse to use an adequate means of contraception (including male patients).
15. Other patients evaluated to be inadequate to participate in the study by co-investigators.
16. No informed consent for either treatment regimen or collection of fresh frozen biopsy tissue for translational studies.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-02; Primary Completion 2014-12 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Fom the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented

SECONDARY OUTCOMES:
Progression free survival (PFS) | Time from registration until objective tumor progression or death for any reason that occurs by the end of the study.
Overall survival (OS) | Time from registration to the date of death.
Time to Treatment Failure (TTF) | Time from registration until discontinuation of treatment for any reason (including progression of disease, treatment toxicity, and death).
Clinical Benefit Rate (CBR) | proportion of patients with confirmed CR, PR, and SD over 24 weeks.
Duration of Response (DR) | Time from first assessment of CR or PR until the first date of PD or death within 60 days of the last tumor assessment or registration, whichever is first.
  Median time will be estimated using the Kaplan Meier method. 95% confidence interval of the median time will be estimated.
Safety Evaluations | Focus on AEs and laboratory assessments.
  AEs will be coded according to the Medical Dictionary for Regulatory Activities Terminology (MedDRA) and the severity of the toxicities will be graded according to the NCI CTCAE criteria, version 3.0, where applicable. Concomitant medications will be coded according to WHO Medication Dictionary for Concomitant Medication.
  All AEs will be summarized (incidence) and listed by the System Organ Class (SOC), preferred term, toxicity/severity grade, and causal relationship. In addition, separate summaries of SAEs and Grade 3 or 4 AEs will be presented. Cardiac AEs including asymptomatic LVEF drops will also be summarized in separate tables.
  Hematological and chemistry laboratory parameters will be graded according to the NCI CTCAE criteria, where applicable. Absolute values and changes from baseline will be summarized by cycle. In addition, worst severity grade will also be summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Peng Yong, MRCP, MB ChB, Principal Investigator — National University Hospital Singapore, NUHS
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore

REFERENCES:
- [Background] Coussens L, Yang-Feng TL, Liao YC, Chen E, Gray A, McGrath J, Seeburg PH, Libermann TA, Schlessinger J, Francke U, et al. Tyrosine kinase receptor with extensive homology to EGF receptor shares chromosomal location with neu oncogene. Science. 1985 Dec 6;230(4730):1132-9. doi: 10.1126/science.2999974.
- [Background] Press MF, Pike MC, Chazin VR, Hung G, Udove JA, Markowicz M, Danyluk J, Godolphin W, Sliwkowski M, Akita R, et al. Her-2/neu expression in node-negative breast cancer: direct tissue quantitation by computerized image analysis and association of overexpression with increased risk of recurrent disease. Cancer Res. 1993 Oct 15;53(20):4960-70. PMID 8104689